CLINICAL TRIAL: NCT04635098
Title: The Effect of Dexmedetomidine on Patients With Chronic Insomnia and Its Influence on Circadian Rhythm:Randomized Clinical Trial, Double Blind
Brief Title: DexmedetOmidine Complement Treats Chronic insOmnia and Improves Circadian Rhythm (DOCTOR)
Acronym: DOCTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOCTOR-super LuoMa
Record Dates: First submitted 2020-11-03; First posted 2020-11-18 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-03

CONDITIONS: Chronic Insomnia
Keywords: Chronic insomnia; Dexmedetomidine; Circadian Rhythm; Sleep monitoring; Brain functional connectivity
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine (Experimental): 0.5μg/kg bolus injection in 10 minutes followed by 0.1µg/kg/hr pump infusion from 23:30 pm to 6:30 am
  Interventions: Drug: dexmedetomidine
- saline (Placebo Comparator): the same rate as dexmedetomidine
  Interventions: Drug: saline

INTERVENTIONS:
Drug: dexmedetomidine — All participants will be randomly assigned to receive either dexmedetomidine or saline
  Other Names: dexmedetomidine group
  Arms: dexmedetomidine
Drug: saline — All participants will be randomly assigned to receive either dexmedetomidine or saline
  Other Names: Placebo group
  Arms: saline

SUMMARY:
It has been reported that dexmedetomidine, alpha-2 adrenoceptor agonist, can activate endogenous neural sleep pathways in the central nervous system. This randomised, double-blinded and controlled trial was designed to investigate whether dexmedetomidine can improve/treat chronic insomnia patients. Its effects on sleep quality and improvement, EEG and circadian rhythm, brain connectivity, cognition and biomarker changes are determined.

DETAILED DESCRIPTION:
Insomnia is a common sleep disorder characterized by difficulty in starting or maintaining sleep, or poor sleep quality and shortened sleep time. The prevalence of insomnia is about 10-20% of population worldwide; Of which about approximately 50% are chronic. Insomnia is a risk factor for cognitive impairment and mental disorder development, and other diseases. Non-pharmacological interventions, e.g. physio-therapy, are often ineffective. Benzodiazepines and their derivatives are commonly prescribed for those patients but their side effects and long-time residual sleepy actions are very risky.

Dexmedetomidine is a highly selective α2 adrenergic receptor agonist with sedative, analgesic and anti-anxiety effects together with remarkable cytoprotective effects. It is widely used as a sedative. Dexmedetomidine was reported promote sleep. It can also modulate "clock" protein expression and hence afford a regulatory effects on the circadian rhythm. This randomised, double-blinded and controlled trial was designed to investigate whether dexmedetomidine can treat chronic insomnia patients. Its effects on sleep quality and improvement, EEG and circadian rhythm, brain connectivity, cognition and biomarker changes are determined. All participants are randomly assigned to receive either dexmedetomidine (a 0.5μg/kg bolus injection for 10 minutes followed by 0.1µg/kg/hr) or placebo (normal saline infusion with an identical protocol as Dex) for 8 hrs from 10pm to 6 am.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18- 65 years old
* Body mass index (BMI) between 18 and 35 kg/m^2；
* Clinical diagnosis of chronic insomnia；
* Must be able to communicate with site personnel

Exclusion Criteria:

* Clinical diagnosis of mental disorders;
* Pregnancy;
* Current use of psychotropic drug ;
* Clinical diagnosis of neurological diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency | Seven hours from day 0 23:30 to day 1 06:30
  measured by polysomnography, Effective sleep time (the sum of non-rapid Eye movement sleep and rapid eye movement sleep time) as a percentage of the monitoring time. Monitoring time is eight hours

SECONDARY OUTCOMES:
BMAL1 | Day 0,Day 1
  sleep protein , Collected from blood lymphocytes
Brain functional connectivity | Seven hours from day 0 23:30 to day 1 06:30
  According to the collected scalp EEG frequency domain and time domain data, the coherence method is used to measure the phase synchronization degree of different brain regions
Interleukin-6(IL-6) | Day 0,Day 1
  cytokines，Collected from blood
Brain-derived neurotrophic factor(BDNF) | Day 0,Day 1
  Collected from blood
N2 sleep time percentage | Seven hours from day 0 23:30 to day 1 06:30
  measured by polysomnography，N2 sleep time as a percentage of total monitoring time. Monitoring time is eight hours
Deep brain functional connectivity | Day 0 before 22:00 , Day 3
  we will analysis the brain connection network according to the functional magnetic resonance imaging nonlinear Granger predictive analysis (Granger causality analysis, GCA) method
Cortisol | Day 0,Day 1
  Collected from blood
Proteomic analysis | Day 0
  Due to some patients having a good response to Dex treatment, while others had rather limited efficacy, we further investigated the proteomic differences in peripheral blood between effective and ineffective patients before their treatment.Screening differential proteins between two groups in the protein database through proteomic analysis results in peripheral blood samples
Sleep latency | Seven hours from day 0 23:30 to day 1 06:30
  measured by polysomnography，the time required from getting ready to go to bed to actually falling asleep
Arousal | Seven hours from day 0 23:30 to day 1 06:30
  measured by polysomnography including arousal > 15 sec(times), micro arousal(times) and wake duration after sleep onset(min).These indicators are used to evaluate the number of awakenings during sleep and the total duration of awakenings.
Sleep diary (sleep duration,sleep latency,arousal) | Day 1,Day 2,Day 3,Day 4,Day 5,Day 6,Day 7
  for one week after treatment recorded by the subjects themselves
Pittsburgh Sleep Quality Index | Day0,Day7
  Scale to assess sleep quality，the lower the score, the better the sleep quality.The minimum value is 0 points, and the maximum value is 21 points.
Insomnia severity index | Day0,Day7
  Scale to assess severity of insomnia,the higher the score, the more severe the insomnia will be.The minimum value is 0 points, and the maximum value is 28 points.
Epworth sleeping scale | Day0,Day7
  A scale for evaluating daytime sleepiness, with higher scores indicating greater daytime sleepiness in subjects.The minimum value is 0 points, and the maximum value is 24 points.
Hamilton anxiety scale | Day0,Day7
  A scale for assessing anxiety levels, where the higher the score, the more anxious the subject is.daytime sleepiness in subjects.The minimum value is 0 points, and the maximum value is 56 points.
Hamilton depression scale | Day0,Day7
  A scale for assessing the degree of depression, with higher scores indicating greater depression among participants.
  0-7 points: No depressive symptoms or normal level; 8-13 points: Mild depressive symptoms; 14-18 points: moderate depressive symptoms; 19-22 points: symptoms of moderate to severe depression; 23 points or above: severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication.No end date.
Access Criteria: Anyone who wishes to access the data for any research purpose.They can get all of the individual participant data collected during the trial, after deidentification.Proposals should be directed to d.ma@imperial.ac.uk/yqz12471@rjh.com.cn.To gain access, data requestors will need to sign a data access agreement. Proteomics data will be available at a website(iprox) following publication.

REFERENCES:
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Akeju O, Hobbs LE, Gao L, Burns SM, Pavone KJ, Plummer GS, Walsh EC, Houle TT, Kim SE, Bianchi MT, Ellenbogen JM, Brown EN. Dexmedetomidine promotes biomimetic non-rapid eye movement stage 3 sleep in humans: A pilot study. Clin Neurophysiol. 2018 Jan;129(1):69-78. doi: 10.1016/j.clinph.2017.10.005. Epub 2017 Oct 20. PMID 29154132